CLINICAL TRIAL: NCT02829229
Title: Community-based Obesity Treatment in African American Women After Childbirth: a Randomized Controlled Trial of Women Infant Children (WIC) Mothers
Brief Title: Community-based Obesity Treatment in African American Women After Childbirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23187; R01HL130816 (NIH)
Record Dates: First submitted 2016-01-28; First posted 2016-07-12 (Estimated); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (UC) (No Intervention): Usual postpartum WIC care
- Community-based obesity treatment (PP) (Experimental): The PP arm includes expanded obesogenic behavior change goals, tailored skills training materials, interactive self-monitoring text messages, video testimonials, and interpersonal counseling support through health coach calls and Facebook.
  Interventions: Behavioral: Community-based obesity treatment (PP)

INTERVENTIONS:
Behavioral: Community-based obesity treatment (PP) — Participants in the treatment (PP) arm will receive a 5-component intervention: 1)Behavior change goals; 2)Self-monitoring; 3)Tailored skills training; 4)Video testimonials & 5)Interpersonal counseling. Both treatment and usual care arms will receive the current standard of care offered to postpartum mothers at WIC.
  Arms: Community-based obesity treatment (PP)

SUMMARY:
The purpose of this study is to determine the effect of the community-based obesity treatment (PP), compared to usual care (UC), on changes in maternal weight over 12 months.

DETAILED DESCRIPTION:
The investigators propose to randomize overweight or obese, African American postpartum WIC participants (n=300) to either usual care (UC) or a community-based obesity treatment (PP) arm. Recruitment will occur in 6 of Philadelphia Women Infants Children's (WIC) clinic sites in the early postpartum period (≤ 6 months after birth). Once enrolled, participants will complete surveys and baseline assessments of their weight, waist circumference, blood pressure, and height at The Center for Obesity Research and Education (CORE). Participants will also have a fasting blood sample taken. Study staff will administer a number of questionnaires assessing demographics, psychosocial factors, contextual factors, and behavioral targets via questionnaires prior to randomization. Participants will then be randomized to the 12-month postpartum weight loss intervention (PP) or usual care (UC). Additional assessments will be conducted at 6 and 12 months post baseline. The PP arm includes expanded obesogenic behavior change goals, tailored skills training materials, interactive self-monitoring text messages, video testimonials, and interpersonal counseling support through health coach calls and Facebook. Data will be analyzed using an intent-to-treat (ITT) approach where subjects are analyzed according to their treatment assignment at randomization, regardless of level of engagement. The primary outcome is weight loss at 12 months. If successful, the expected results could provide a sustainable, low-cost, postpartum weight loss intervention model for widespread dissemination to reduce disparities in obesity and cardiometabolic comorbidities.

ELIGIBILITY:
Inclusion Criteria:

1. Self-identification as African American
2. Self-report pre-pregnancy BMI between 25-49.9 kg/m2
3. Measured BMI at baseline between 25-49.9 kg/m2
4. Philadelphia WIC participant
5. Singleton birth
6. Between 1 and 6 months postpartum
7. Own a cell phone with an unlimited text messaging plan
8. Able to participate in light physical activity (walking)
9. Participants must be willing to comply with all study-related procedures
10. Participants must be able to read and write fluently in English

Exclusion Criteria:

1. BMI ≤ 24.9 or ≥ 50.0 kg/m2
2. Uncontrolled hypertension (systolic blood pressure > 160 or diastolic blood pressure > 95 mmHg). Participants with controlled hypertension on medication for at least three months are allowable.
3. Known atherosclerotic cardiovascular disease
4. Known congestive heart failure
5. Known diabetes mellitus (type 1 or type 2)
6. Known thyroid disease
7. Any major active rheumatologic, pulmonary, hepatic, dermatologic disease or inflammatory condition requiring steroids or immune modulating medications
8. History of testing HIV positive
9. Current smoker or tobacco user. Participants with < 5 cigarettes daily are allowable
10. Current or recent history (past 6 months) of drug or alcohol abuse or dependence
11. Participation in any weight control or investigational drug study within 6 weeks of screening
12. Current consumption of any of the following medications: appetite suppressants, anti-psychotics, lipase inhibitors
13. Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety for successful participation in the study
14. Gastrointestinal Disorders (gallbladder disease, Crohn's disease, etc)
15. Previous weight loss surgery
16. History of bulimia or anorexia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Weight loss (kilograms) | At baseline and 12 months
  Weight will be measured using a calibrated scale at baseline and 12-month follow-up. Weight loss will be calculated as the difference between mean 12-month and baseline weight in kilograms.

SECONDARY OUTCOMES:
Obesogenic dietary behaviors | At baseline and 12 months
  Using National Cancer Institute's Diet History Questionnaire, the investigators will assess categories of sugary drink intake, fast/fried food intake, and snacking at baseline and 12-month follow-up.
Insulin Resistance | At baseline and 12 months
  Blood will be drawn to assess insulin resistance (insulin and glucose). The Homeostatic model assessment for Insulin Resistance (HOMA-IR) calculation will be used to quantify participant mean insulin resistance at baseline and 12-month follow-up.
Health-related quality of life | At baseline and 12 months
  Short Form-12 (SF-12) questionnaire will be used to collect health-related quality of life at baseline and 12-month follow-up.
Physical Activity | At baseline and 12 months
  Wrist Actigraphy will be used to measure physical activity (average number of steps) at baseline and 12-month follow-up.
Physical Activity | At baseline and 12 months
  Wrist Actigraphy will be used to measure physical activity (average intensity of activity) at baseline and 12-month follow-up.
Sleep | At baseline and 12 months
  Wrist Actigraphy will be used to measure sleep (mean duration of sleep) at baseline and 12-month follow-up.
Sleep | At baseline and 12 months
  Wrist Actigraphy will be used to measure sleep (mean sleep efficiency) at baseline and 12-month follow-up.
Sleep | At baseline and 12 months
  Wrist Actigraphy will be used to measure sleep (mean wake after sleep onset) at baseline and 12-month follow-up.
Hemoglobin A1c (HbA1c) | At baseline and 12 months
  Hemoglobin A1c test will be performed by a lab to identify the 3-month average plasma glucose concentration at baseline and 12-month follow-up. The investigators will categorize participants as no diabetes (HbA1c <5.7), prediabetes (HBA1c 5.7-6.4), and diabetes (HBA1c >6.4) at both timepoints.
Lipids | At baseline and 12 months
  Total cholesterol test will be performed by a lab to identify mean total blood cholesterol level, low density lipoprotein and high density lipoprotein levels at baseline and 12-month follow-up.

OTHER OUTCOMES:
Utilize Reach Effectiveness Adoption Implementation (RE-AIM) to evaluate the intervention's dissemination potential | 12 months
  The five steps are Reach the target population; Effectiveness; Adoption by target staff, settings or institutions; Implementation consistency, costs and adaptions made during delivery and Maintenance of intervention effects in individuals and settings over time. Previously collected data such as target population characteristics; attrition and completion percentages; results related to primary, secondary and unintended outcomes; intervention fidelity; participant knowledge application and sustainability will be used within scope of 5 steps to determine dissemination potential.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon J Herring, MD MPH, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Dr. Herring (PI) will ensure that all publications that result from data collected as part of this project will comply with the NIH public access policy. Also, Dr. Herring agrees to develop a transportable de-identified database, codebook, and mechanism by which data can be shared with other investigators upon approval of the study's research team. The Resource Sharing Plan will be reviewed and approved by Temple University's Institutional Review Board.